CLINICAL TRIAL: NCT03678883
Title: Phase 1/2 Study of 9-ING-41, a Glycogen Synthase Kinase-3 Beta (GSK-3β) Inhibitor, As a Single Agent and Combined with Chemotherapy, in Patients with Refractory Hematologic Malignancies or Solid Tumors
Brief Title: 9-ING-41 in Patients with Advanced Cancers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Actuate Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1801
Record Dates: First submitted 2018-09-15; First posted 2018-09-20 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Pancreatic Cancer; Sarcoma; Renal Cancer; Refractory Cancer; Refractory Neoplasm; Refractory Non-Hodgkin Lymphoma; Pancreatic Adenocarcinoma; Resistant Cancer; Neoplasm Metastasis; Neoplasm of Bone; Neoplasm, Breast; Neoplasm of Lung; Neoplasms,Colorectal; Neoplasms Pancreatic; Malignant Glioma; Malignancies; Malignancies Multiple; Bone Metastases; Bone Neoplasm; Bone Cancer; Pancreas Cancer; Pancreatic Neoplasms; Breast Neoplasms; Acute T Cell Leukemia Lymphoma
Keywords: Refractory cancers; 9-ING-41; Glycogen Synthase Kinase; GSK-3β; NF-κβ; Apoptosis; Chemoresistance; DNA damage response DDR; Ataxia telangiectasia mutated and Rad3 related ATR; Checkpoint kinase 1 CHK1; Checkpoint Inhibitor; LAG-3; ATLL
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Sarcoma; Kidney Neoplasms; Lymphoma, Non-Hodgkin; Neoplasm Metastasis; Bone Neoplasms; Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Glioma; Hereditary Sensory and Autonomic Neuropathies; Leukemia-Lymphoma, Adult T-Cell | interventions — 3-(5-fluorobenzofuran-3-yl)-4-(5-methyl-5H-(1,3)dioxolo(4,5-f)indol-7-yl)-pyrrole-2,5-dione; Gemcitabine; Doxorubicin; liposomal doxorubicin; Lomustine; Carboplatin; Taxes; Albumin-Bound Paclitaxel; Paclitaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- 9-ING-41 (Experimental): Drug: 9-ING-41
  Interventions: Drug: 9-ING-41
- 9-ING-41 plus Gemcitabine (Experimental): Drugs: Gemcitabine - 21 day cycle. 9-ING-41
  Interventions: Drug: 9-ING-41; Drug: Gemcitabine - 21 day cycle
- 9-ING-41 plus Doxorubicin (Experimental): Drugs: Doxorubicin. 9-ING-41
  Interventions: Drug: 9-ING-41; Drug: Doxorubicin.
- 9-ING-41 plus Lomustine (Experimental): Drugs: Lomustine. 9-ING-41.
  Interventions: Drug: 9-ING-41; Drug: Lomustine
- 9-ING-41 plus Carboplatin (Experimental): Drugs: Carboplatin. 9-ING-41.
  Interventions: Drug: 9-ING-41; Drug: Carboplatin.
- 9-ING-41 plus nab paclitaxel Gemcitabine (Experimental): Drugs: Nab-paclitaxel. Gemcitabine - 28 day cycle. 9-ING-41.
  Interventions: Drug: 9-ING-41; Drug: Nab paclitaxel.; Drug: Gemcitabine - 28 day cycle
- 9-ING-41 plus Paclitaxel/Carboplatin (Experimental): Drugs: Paclitaxel. Carboplatin. 9-ING-41.
  Interventions: Drug: 9-ING-41; Drug: Carboplatin.; Drug: Paclitaxel.
- 9-ING-41 plus Irinotecan (Experimental): Drugs: Irinotecan. 9-ING-41.
  Interventions: Drug: 9-ING-41; Drug: Irinotecan

INTERVENTIONS:
Drug: 9-ING-41 — Starting dose of-9-ING-41 will be administered on Day 1 and 4 each week of a 21-day cycle. 9-ING-41 will be administered intravenously over 60 minutes.
Drug: Gemcitabine - 21 day cycle — Gemcitabine 1250 mg/m2 as a 30-minute intravenous infusion on Days 1 and 8 of a 21-day cycle
  Other Names: Gemzar
  Arms: 9-ING-41 plus Gemcitabine
Drug: Doxorubicin. — Doxorubicin 75 mg/m2, intravenous bolus on Day 1 of a 21-day cycle up to a maximum lifetime dose of 550 mg/m2.
  Other Names: Doxil; Adriamycin
  Arms: 9-ING-41 plus Doxorubicin
Drug: Lomustine — Lomustine 30 mg/m² orally as a single dose, weekly for twelve weeks.
  Other Names: CCNU; Gleostine
  Arms: 9-ING-41 plus Lomustine
Drug: Carboplatin. — Carboplatin AUC 6 IV over 1 hour on Day 1 of a 21-day cycle.
  Other Names: Paraplatin
  Arms: 9-ING-41 plus Carboplatin; 9-ING-41 plus Paclitaxel/Carboplatin
Drug: Nab paclitaxel. — Nab-paclitaxel 125 mg/m2 intravenously on Days 1, 8 and 15 of a 28-day cycle
  Other Names: Abraxane; Protein-bound paclitaxel; Nanoparticle albumin-bound paclitaxel
  Arms: 9-ING-41 plus nab paclitaxel Gemcitabine
Drug: Paclitaxel. — Paclitaxel 175 mg/m2 intravenously over 3 hours on Day 1 of a 21-day cycle.
  Other Names: Taxol
  Arms: 9-ING-41 plus Paclitaxel/Carboplatin
Drug: Gemcitabine - 28 day cycle — Gemcitabine 1000 mg/m2 intravenously over 30-minutes on Days 1, 8 and 15 of a 28-day cycle
  Other Names: Gemzar
  Arms: 9-ING-41 plus nab paclitaxel Gemcitabine
Drug: Irinotecan — Irinotecan 350 mg/m2 intravenously over 90-minutes on Day 1 of a 21-day cycle
  Other Names: Camptosar
  Arms: 9-ING-41 plus Irinotecan

SUMMARY:
GSK-3β is a potentially important therapeutic target in human malignancies. The Actuate 1801 Phase 1/2 study is designed to evaluate the safety and efficacy of 9-ING-41, a potent GSK-3β inhibitor, as a single agent and in combination with cytotoxic agents, in patients with refractory cancers.

DETAILED DESCRIPTION:
9-ING-41 is a first-in-class, intravenously administered, maleimide-based small molecule potent selective GSK-3β inhibitor with significant pre-clinical antitumor activity. GSK-3 is a serine/threonine kinase initially described as a key regulator of metabolism and has a role in diverse disease processes including cancer, immune disorders, pathologic fibrosis, metabolic disorders, and neurological disorders. GSK-3 has two ubiquitously expressed and highly conserved isoforms, GSK-3α and GSK-3β, with both shared and distinct substrates and functional effects. GSK-3β is particularly important in tumor progression and modulation of oncogenes (including beta-catenin, cyclin D1 and c-Myc), cell cycle regulators (e.g. p27Kip1) and mediators of epithelial-mesenchymal transition (e.g. zinc finger protein SNAI1, Snail). Aberrant overexpression of GSK-3β has been shown to promote tumor growth and chemotherapy resistance in various solid tumors including colon, ovarian, and pancreatic cancers and glioblastoma through differential effects on the pro-survival nuclear factor kappa-light-chain-enhancer of activated B cells (NF-κB) and c-Myc pathways as well on tumor necrosis factor-related apoptosis-inducing ligand (TRAIL) and p53-mediated apoptotic mechanisms. GSK-3β helps maintain malignant cell survival and proliferation, particularly in terms of mediating resistance to standard anti-cancer therapies, through the NF-κB pathway. GSK-3β has been established as a potential anticancer target in human bladder, breast, colorectal, glioblastoma, lung, neuroblastoma, ovarian, pancreatic, prostate, renal and thyroid cancers as well as chronic lymphocytic leukemia and lymphomas.

9-ING-41 is a small molecule potent selective GSK-3β inhibitor with broad spectrum pre-clinical antitumor activity. It's modes of action include downregulation of NF-κB and decreasing the expression NF-κB target genes including cyclin D1, Bcl-2, anti-apoptotic protein (XIAP) and B-cell lymphoma-extra large (Bcl-XL) leading to inhibition of tumor growth in multiple solid tumor cell and lymphoma lines and patient derived xenograft (PDX) models. NF-κB is constitutively active in cancer cells and promotes anti-apoptotic molecule expression. NF-κB activation is particularly important in cancer cells that have become chemo- and/or radio-resistant. 9-ING-41 also has significant activity in pre-clinical models of pathological pleural and pulmonary fibrosis. 9-ING-41 has significant in vitro and in vivo activity as a single agent and/or in combination with standard cytotoxic chemotherapies in a spectrum of solid tumors and hematological malignancies including bladder, breast, glioblastoma, neuroblastoma, pancreatic, sarcomas, and renal cancers as well as lymphomas.

The 1801 had three parts:

* Completed: Part 1 (9-ING-41 as monotherapy): The standard 3+3 dose escalation design will be applied to all dose cohorts until the Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) is identified.
* Completed: 9-ING-41 combined with standard anticancer agents: The 3+3 dose escalation study design will be used for 8 chemotherapy combination regimens (9-ING-41 plus gemcitabine, doxorubicin, lomustine, carboplatin, irinotecan, nab-paclitaxel plus gemcitabine, paclitaxel plus carboplatin, pemetrexed plus carboplatin) to identify the MTD/RP2D of each regimen.
* Part 3: A randomized Phase 2 study of 9-ING-41 either once or twice weekly with gemcitabine and nab-paclitaxel (GA) versus GA alone for patients with previously untreated metastatic or locally advanced pancreatic cancer is now open.

ELIGIBILITY:
Inclusion Criteria:

* Patient -

  1. Is able to understand and voluntarily sign a written informed consent and is willing and able to comply with the protocol requirements including scheduled visits, treatment plan, laboratory tests and other study procedures.
  2. Is aged ≥ 18 years
  3. Has pathologically confirmed advanced or metastatic malignancy characterized by one or more of the following:

     1. Patient is intolerant of existing therapy(ies) known to provide clinical benefit for their condition
     2. Malignancy is refractory to existing therapy(ies) known to potentially provide clinical benefit
     3. Malignancy has relapsed after standard therapy
     4. Malignancy for which there is no standard therapy that improves survival by at least 3 months
  4. Has evaluable tumor(s) by standard radiological and/or laboratory assessments as applicable to their malignancy - in Part 3, patients with solid tumors must have least 1 measurable lesion per response evaluation criteria in solid tumors (RECIST) v1.1 criteria, measured preferably by computed tomography (CT) scan or magnetic resonance image (MRI). In the case of patients with glioblastoma multiforme (GBM) or other central nervous system (CNS) tumors, the tumor must be measurable, defined as a clearly enhancing tumor with at two perpendicular diameters at entry equal or superior to 1cm.
  5. Has laboratory function within specified parameters (may be repeated):

     1. Adequate bone marrow function: absolute neutrophil count (ANC) ≥ 500/mL; hemoglobin ≥ 8.5 g/dL, platelets ≥ 50,000/mL
     2. Adequate liver function: transaminases (aspartate aminotransferase/ alanine aminotransferase, AST/ALT) and alkaline phosphatase ≤ 3 (≤ 5 X the upper limit of normal (ULN) in the setting of liver metastasis or infiltration with malignant cells) x ULN; bilirubin ≤ 1.5 x ULN
     3. Adequate renal function: creatinine clearance ≥ 60 mL/min (Cockcroft and Gault)
     4. Adequate blood coagulation: international normalized ratio (INR) ≤ 2.3
     5. Serum amylase and lipase ≤ 1.5 x ULN
  6. Has adequate performance status (PS): Eastern Co-operative Oncology Group (ECOG) PS 0-2
  7. Has received the final dose of any of the following treatments/ procedures with the specified minimum intervals before first dose of study drug (unless in the opinion of the investigator and the study medical coordinator the treatments/ procedures will not compromise patient safety or interfere with study conduct and with IDMC agreement):

     * Chemotherapy, immunotherapy, or systemic radiation therapy - 14 days or ≥ 5 half-lives (whichever is shorter)
     * Focal radiation therapy - 7 days
     * Systemic and topical corticosteroids - 7 days
     * Surgery with general anesthesia - 7 days
     * Surgery with local anesthesia - 3 days
  8. May continue endocrine therapies (e.g. for breast or prostate cancer) and/or anti-human epidermal growth factor (Her2) therapies while on this study
  9. Women of childbearing potential must have a negative baseline blood or urine pregnancy test within 72 hours of first study therapy. Women may be neither breastfeeding nor intending to become pregnant during study participation and must agree to use effective contraceptive methods (hormonal or barrier method of birth control, or true abstinence) for the duration of study participation and in the following 90 days after discontinuation of study treatment
  10. Male patients with partners of childbearing potential must take appropriate precautions to avoid fathering a child from screening until 90 days after discontinuation of study treatment and use appropriate barrier contraception or true abstinence
  11. Must not be receiving any other investigational medicinal product

Exclusion Criteria:

* Patient -

  1. Is pregnant or lactating
  2. Is known to be hypersensitive to any of the components of 9-ING-41 or to the excipients used in its formulation
  3. Has not recovered from clinically significant toxicities as a result of prior anticancer therapy, except alopecia and infertility. Recovery is defined as ≤ Grade 2 CTCAE Version 4.03
  4. Has significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, or stroke within 6 months of the first dose of 9-ING-41, or cardiac arrhythmia requiring medical treatment detected at screening
  5. Has had a myocardial infarction within 12 weeks of the first dose of 9-ING-41 or has electrocardiogram (ECG) abnormalities that are deemed medically relevant by the investigator or study medical coordinator
  6. Has known symptomatic rapidly progressive brain metastases or leptomeningeal involvement as assessed by CT scan or MRI. Patients with stable asymptomatic brain metastases or leptomeningeal disease or slowly progressive disease are eligible provided that they have not required new treatments for this disease in a 28-day period before the first dose of study drug, and anticonvulsants and steroids are at a stable dose for a period of 14 days prior to the first dose of study drug
  7. Has had major surgery (not including placement of central lines) within 7 days prior to study entry or is planned to have major surgery during the course of the study (major surgery may be defined as any invasive operative procedure in which an extensive resection is performed, e.g. a body cavity is entered, organs are removed, or normal anatomy is altered. In general, if a mesenchymal barrier is opened (pleural cavity, peritoneum, meninges), the surgery is considered major)
  8. Has any medical and/or social condition which, in the opinion of the investigator or study medical coordinator would preclude study participation
  9. Has received an investigational anti-cancer drug in the 14-day period before the first dose of study drug (or within 5 half-lives if longer) or is currently participating in another interventional clinical trial
  10. Has a current active malignancy other than the target cancer
  11. Is considered to be a member of a vulnerable population (for example, prisoners)

Part 3 ARMB Inclusion Criteria: Patient -

1. Is able to understand and voluntarily sign a written informed consent and is willing and able to comply with the protocol requirements including scheduled visits, treatment plan, laboratory tests and other study procedures
2. Is aged ≥ 18 years
3. Has pathologically confirmed metastatic pancreatic cancer AND is previously untreated with systemic agents in the recurrence/metastatic setting.
4. Must have at least 1 measurable lesion per RECIST v1.1, measured preferably by computed tomography (CT) scan or magnetic resonance image (MRI)
5. Has laboratory function within specified parameters (may be repeated):

   e. Adequate bone marrow function: absolute neutrophil count (ANC) ≥ 500/mL; hemoglobin ≥ 8.5 g/dL, platelets ≥ 75,000/mL f. Adequate liver function: transaminases (aspartate aminotransferase/ alanine aminotransferase, AST/ALT) and alkaline phosphatase ≤ 3 (≤ 10 X the upper limit of normal (ULN) in the setting of liver metastasis or infiltration with malignant cells) x ULN; bilirubin ≤ 1.5 x ULN Adequate renal function: creatinine clearance ≥ 30 mL/min (Cockcroft and Gault)
6. Has Eastern Co-operative Oncology Group (ECOG) PS 0 or 1
7. Has received the final dose of any of the following treatments/ procedures with the specified minimum intervals before first dose of study drug:

   * Focal radiation therapy - 7 days
   * Surgery with general anesthesia - 7 days
   * Surgery with local anesthesia - 3 days
8. May have received treatment with fluorouracil or gemcitabine as a radiation sensitizer in the adjuvant setting if the treatment was received at least 6 months before study enrollment
9. May have received neoadjuvant chemotherapy with FOLFIRINOX if last dose given at least 6 months before study enrollment
10. May have received prior cytotoxic doses of systemic chemotherapy in the adjuvant setting if last dose given at least 6 months before study enrollment
11. Women of childbearing potential must have a negative baseline blood or urine pregnancy test within 72 hours of first study therapy. Women may be neither breastfeeding nor intending to become pregnant during study participation and must agree to use effective contraceptive methods (hormonal or barrier method of birth control, or true abstinence) for the duration of study participation and in the following 90 days after discontinuation of study treatment
12. Male patients with partners of childbearing potential must take appropriate precautions to avoid fathering a child from screening until 90 days after discontinuation of study treatment and use appropriate barrier contraception or true abstinence
13. Must not be receiving any other investigational medicinal product

Patient who meets ANY of the following criteria is not eligible for this Part 3 study Arm B:

Exclusion Criteria:

1. Is pregnant or lactating
2. Is known to be hypersensitive to any of the components of 9-ING-41 or to the excipients used in its formulation
3. Has endocrine or acinar pancreatic carcinoma
4. Has not recovered from clinically significant toxicities as a result of prior anticancer therapy, except alopecia and/or infertility. Recovery is defined as ≤ Grade 2 severity per CTCAE, v5.0
5. Has significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, or stroke within 6 months of the first dose of study therapy, or uncontrolled cardiac arrhythmia
6. Has had a myocardial infarction within 12 weeks of the first dose of study therapy or has electrocardiogram (ECG) abnormalities that are deemed medically relevant by the investigator
7. Has symptomatic rapidly progressive brain metastases or leptomeningeal involvement as assessed by CT scan or MRI. Patients with stable brain metastases or leptomeningeal disease or slowly progressive disease are eligible provided that they have not required new treatments for this disease in a 28-day period before the first dose of study drug, and anticonvulsants and steroids are at a stable dose for a period of 14 days prior to the first dose of study drug
8. Has had major surgery (not including placement of central lines) within 7 days prior to study entry or is planned to have major surgery during the course of the study (major surgery may be defined as any invasive operative procedure in which an extensive resection is performed, e.g., a body cavity is entered, organs are removed, or normal anatomy is altered. In general, if a mesenchymal barrier is opened (pleural cavity, peritoneum, meninges), the surgery is considered major)
9. Has any medical and/or social condition which, in the opinion of the investigator or study medical coordinator would preclude study participation.
10. Has received an investigational anti-cancer drug in the 14-day period before the first dose of study drug (or within 5 half-lives if longer) or is currently participating in another interventional clinical trial.
11. Has a current active malignancy other than pancreatic cancer
12. Is considered to be a member of a vulnerable population (for example, prisoners).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Parts 1/2: Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 3 months to 3 years
  The standard assessments used to assign a score to any affected organ system as per the NCI CTCAE 4.03 will be conduced at each protocol-specified timepoint.
Part 3 Arm B | 3 months to 3 years
  To determine the 1-year survival rate of patients treated on the 9-ING-41 schedule chosen from the run-in stage of the study compared to the control arm

CONTACTS AND LOCATIONS:
Locations (66):
- United States (40):
  - Mayo Clinic, Phoenix, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California Irvine Health, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Miami Cancer Institute, Miami, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - Kansas University Cancer Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - MetroMetro-Minnesota Community Oncology Research Consortium (MMCORC), Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - Capital Health Medical Center/ Hopewell, Pennington, New Jersey
  - MD Anderson Cancer Center at Cooper, Voorhees Township, New Jersey
  - Columbia University- Irving Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Sanford Research, Sioux Falls, South Dakota
  - West Cancer Center, Germantown, Tennessee
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Sarah Cannon Research Institute- Tennessee Oncology-Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology- Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - UW Carbone Cancer Center, Madison, Wisconsin
- Belgium (4):
  - UZA- Antwerpen, Edegem, Antwerp
  - Imelda VZW, Bonheiden
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre, Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- France (7):
  - Center Hospitalier Regional Universitaire de Besancon - Site Jean Minjoz, Besançon, Bourgogne-Franche-Comté
  - CHRU Brest Hopital Morvan, Brest, Brittany Region
  - Hopital Claude Huriez, Lille, Hauts-de-France
  - Institute de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Institut Bergonie, Bordeaux, Nouvelle-Aquitaine
  - Insitut de Cancerologie de l'Ouest, Saint-Herblain, Pays de la Loire Region
  - Hopital de la Timone, Marseille
- Netherlands Cancer Institute, Amsterdam, Netherlands
- Portugal (3):
  - Fundacao Champalimaud, Lisbon
  - Hospital Da Luz, Lisbon
  - Centro Hospitalar Universitario Sao Joao, Porto
- Spain (5):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Hospital Clinico U San Carlos (HSC), Madrid
  - START Madrid-HM CIOCC Hospital Universitario, Madrid
  - INCLIVA University of Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ugolkov AV, Bondarenko GI, Dubrovskyi O, Berbegall AP, Navarro S, Noguera R, O'Halloran TV, Hendrix MJ, Giles FJ, Mazar AP. 9-ING-41, a small-molecule glycogen synthase kinase-3 inhibitor, is active in neuroblastoma. Anticancer Drugs. 2018 Sep;29(8):717-724. doi: 10.1097/CAD.0000000000000652. PMID 29846250
- [Background] Karmali R, Chukkapalli V, Gordon LI, Borgia JA, Ugolkov A, Mazar AP, Giles FJ. GSK-3beta inhibitor, 9-ING-41, reduces cell viability and halts proliferation of B-cell lymphoma cell lines as a single agent and in combination with novel agents. Oncotarget. 2017 Nov 11;8(70):114924-114934. doi: 10.18632/oncotarget.22414. eCollection 2017 Dec 29. PMID 29383130
- [Background] Ugolkov A, Qiang W, Bondarenko G, Procissi D, Gaisina I, James CD, Chandler J, Kozikowski A, Gunosewoyo H, O'Halloran T, Raizer J, Mazar AP. Combination Treatment with the GSK-3 Inhibitor 9-ING-41 and CCNU Cures Orthotopic Chemoresistant Glioblastoma in Patient-Derived Xenograft Models. Transl Oncol. 2017 Aug;10(4):669-678. doi: 10.1016/j.tranon.2017.06.003. Epub 2017 Jun 30. PMID 28672195
- [Background] Ugolkov A, Gaisina I, Zhang JS, Billadeau DD, White K, Kozikowski A, Jain S, Cristofanilli M, Giles F, O'Halloran T, Cryns VL, Mazar AP. GSK-3 inhibition overcomes chemoresistance in human breast cancer. Cancer Lett. 2016 Oct 1;380(2):384-392. doi: 10.1016/j.canlet.2016.07.006. Epub 2016 Jul 14. PMID 27424289
- [Background] Pal K, Cao Y, Gaisina IN, Bhattacharya S, Dutta SK, Wang E, Gunosewoyo H, Kozikowski AP, Billadeau DD, Mukhopadhyay D. Inhibition of GSK-3 induces differentiation and impaired glucose metabolism in renal cancer. Mol Cancer Ther. 2014 Feb;13(2):285-96. doi: 10.1158/1535-7163.MCT-13-0681. Epub 2013 Dec 10. PMID 24327518
- [Background] Walz A, Ugolkov A, Chandra S, Kozikowski A, Carneiro BA, O'Halloran TV, Giles FJ, Billadeau DD, Mazar AP. Molecular Pathways: Revisiting Glycogen Synthase Kinase-3beta as a Target for the Treatment of Cancer. Clin Cancer Res. 2017 Apr 15;23(8):1891-1897. doi: 10.1158/1078-0432.CCR-15-2240. Epub 2017 Jan 4. PMID 28053024
- [Background] Ugolkov AV, Matsangou M, Taxter TJ, O'Halloran TV, Cryns VL, Giles FJ, Mazar AP. Aberrant expression of glycogen synthase kinase-3beta in human breast and head and neck cancer. Oncol Lett. 2018 Nov;16(5):6437-6444. doi: 10.3892/ol.2018.9483. Epub 2018 Sep 21. PMID 30405781
- [Background] Sahin I, Eturi A, De Souza A, Pamarthy S, Tavora F, Giles FJ, Carneiro BA. Glycogen synthase kinase-3 beta inhibitors as novel cancer treatments and modulators of antitumor immune responses. Cancer Biol Ther. 2019;20(8):1047-1056. doi: 10.1080/15384047.2019.1595283. Epub 2019 Apr 12. PMID 30975030
- [Background] Wu X, Stenson M, Abeykoon J, Nowakowski K, Zhang L, Lawson J, Wellik L, Li Y, Krull J, Wenzl K, Novak AJ, Ansell SM, Bishop GA, Billadeau DD, Peng KW, Giles F, Schmitt DM, Witzig TE. Targeting glycogen synthase kinase 3 for therapeutic benefit in lymphoma. Blood. 2019 Jul 25;134(4):363-373. doi: 10.1182/blood.2018874560. Epub 2019 May 17. PMID 31101621
- [Background] Ding L, Madamsetty VS, Kiers S, Alekhina O, Ugolkov A, Dube J, Zhang Y, Zhang JS, Wang E, Dutta SK, Schmitt DM, Giles FJ, Kozikowski AP, Mazar AP, Mukhopadhyay D, Billadeau DD. Glycogen Synthase Kinase-3 Inhibition Sensitizes Pancreatic Cancer Cells to Chemotherapy by Abrogating the TopBP1/ATR-Mediated DNA Damage Response. Clin Cancer Res. 2019 Nov 1;25(21):6452-6462. doi: 10.1158/1078-0432.CCR-19-0799. Epub 2019 Sep 18. PMID 31533931
- [Background] Jeffers A, Qin W, Owens S, Koenig KB, Komatsu S, Giles FJ, Schmitt DM, Idell S, Tucker TA. Glycogen Synthase Kinase-3beta Inhibition with 9-ING-41 Attenuates the Progression of Pulmonary Fibrosis. Sci Rep. 2019 Dec 12;9(1):18925. doi: 10.1038/s41598-019-55176-w. PMID 31831767
- [Background] Kuroki H, Anraku T, Kazama A, Bilim V, Tasaki M, Schmitt D, Mazar AP, Giles FJ, Ugolkov A, Tomita Y. 9-ING-41, a small molecule inhibitor of GSK-3beta, potentiates the effects of anticancer therapeutics in bladder cancer. Sci Rep. 2019 Dec 27;9(1):19977. doi: 10.1038/s41598-019-56461-4. PMID 31882719
- [Background] Anraku T, Kuroki H, Kazama A, Bilim V, Tasaki M, Schmitt D, Mazar A, Giles FJ, Ugolkov A, Tomita Y. Clinically relevant GSK-3beta inhibitor 9-ING-41 is active as a single agent and in combination with other antitumor therapies in human renal cancer. Int J Mol Med. 2020 Feb;45(2):315-323. doi: 10.3892/ijmm.2019.4427. Epub 2019 Dec 12. PMID 31894292
- [Derived] Hsu A, Huntington KE, De Souza A, Zhou L, Olszewski AJ, Makwana NP, Treaba DO, Cavalcante L, Giles FJ, Safran H, El-Deiry WS, Carneiro BA. Clinical activity of 9-ING-41, a small molecule selective glycogen synthase kinase-3 beta (GSK-3beta) inhibitor, in refractory adult T-Cell leukemia/lymphoma. Cancer Biol Ther. 2022 Dec 31;23(1):417-423. doi: 10.1080/15384047.2022.2088984. PMID 35815408
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903